CLINICAL TRIAL: NCT06071416
Title: The Lateral Approach Maxillary Sinus Floor Augmentation Using Biphasic Material Combined With Injectable Platelet Rich Fibrin- Randomized Clinical Trial
Brief Title: Biphasic Material With PRF in Lateral Sinus Floor Augmentation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alzahraa Alghriany, Lecturer, Oral medicine, Periodontology and Oral diagnosis, Faculty of dentistry, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRF in sinus augmentation
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Maxillary Sinus Disease
Keywords: sinus floor augmentation; biphasic calcium phosphate; PRF
MeSH Terms: interventions — hydroxyapatite-beta tricalcium phosphate

STUDY DESIGN:
Intervention Model Description: Group I, patients undergo sinus lifting using bone substitute BCP alone.
  -Group II, patients who undergo sinus lifting using BCP with I-PRF.
Who Masked: Participant, Outcomes Assessor
Masking Description: using automated sequence generation ( randomizer. org) patients will be divided into the two groups ,In sequentially numbered , opaque, sealed envelopes, participants will be enrolled and evaluated while the allocation sequence will be kept a secret from the researchers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 BCP alone (Active Comparator): Lateral bone augmentation with biphasic calcium phosphate BCP bone substitute application
  Interventions: Procedure: Lateral sinus floor augmentation; Drug: Biphasic Calcium Phosphate
- Group 2 BCP with I-PRF (Active Comparator): Lateral bone augmentation with biphasic calcium phosphate BCP bone substitute application with addition of injectable platlet rich fibrin I-PRF
  Interventions: Procedure: Lateral sinus floor augmentation; Drug: Biphasic Calcium Phosphate; Procedure: Injectable platlets rich fibrin

INTERVENTIONS:
Procedure: Lateral sinus floor augmentation — maxillary sinus floor augmentation by lateral approach
Drug: Biphasic Calcium Phosphate — appliaction of BCP bone substitute
Procedure: Injectable platlets rich fibrin — centrifuge 10 ml of patient blood to get I-PRF that applied to the bone substitute
  Arms: Group 2 BCP with I-PRF

SUMMARY:
A lack of bone in the posterior maxilla, mainly resulting from the combination of alveolar bone resorption after tooth loss, pneumatization of the maxillary sinus, and periodontal disease, leads to increased difficulty during dental implant treatment.

The classic technique for maxillary sinus floor augmentation entails the preparation of the trap door to elevate the schneiderian membrane in the lateral sinus wall. it can be done either in a single stage with simultaneous implant placement or in two stages with delayed implant placement, depending on the available residual alveolar ridge height that necessary for implant primary stability.

The new compartment created between the floor of maxillary sinus and the elevated membrane was filled with either autogenous, allografts, xenograft or combination of them to maintain space for new bone formation. The disadvantages of such methods are high costs for grafting material, time consuming and high morbidity, because harvesting of bone grafts is needed.

DETAILED DESCRIPTION:
Recently, a systematic review demonstrated the effectiveness of synthetic bone materials, including biphasic calcium phosphate (BCP), as substitutes for autogenous bone. BCP consists of hydroxyapatite (HA) and β-tricalcium phosphate (β-TCP). In contrast with stable HA, β-TCP is highly resorptive and is replaced by newly formed bone; therefore, the resorption rate of BCP could be influenced by the ratio of HA and β-TCP.

platelet-rich fibrin (PRF) was recently introduced as additional or replacement materials in bone augmentation procedures. The use of biologic mediators with osteoinductive properties has been considered to reduce the time interval and accelerate the formation of new bone. The strengths of PRF in reducing tissue inflammation, promoting the vascularization of bone tissue, accelerating new bone formation, and improving scaffold mechanics have been reported.

ELIGIBILITY:
Inclusion Criteria:

* Residual bone crest height < 5 mm and width≥6 mm in the planned implant site.
* Healed bone crest (at least 6 months elapsed from tooth loss/extraction);

Exclusion Criteria:

* Absolute medical contraindications to implant surgery such as uncontrolled diabetes mellitus, blood platelet disorders, serious osseous disorders, and cardiac arrhythmia; history of bone grafting in the posterior maxilla, immunocompromised patients, taking corticosteroids, taking aspirin before the procedure, positive history of chemotherapy and radiotherapy, and maxillary sinus pathologies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Vertical bone gain BG | 6 months
  Vertical bone gain (BG) 6 months after sinus augmentation in both height and density aspects by cone beam CT

IPD SHARING:
Plan to Share IPD: No